CLINICAL TRIAL: NCT00741364
Title: Randomized Trial of the Effects of Vitamin D on Prostate Cancer-associated Lesions and on Vitamin D Metabolites in Prostate
Brief Title: Vitamin D Effects on Prostate Pathology
Acronym: DProstate
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Toronto (Other)
Collaborators: Mount Sinai Hospital, Canada (Other); University Health Network, Toronto (Other); Sunnybrook Health Sciences Centre (Other); Canadian Cancer Society (CCS) (Other)
Responsible Party: Principal Investigator, Reinhold Vieth, Dr. Reinhold Vieth, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M2140
Record Dates: First submitted 2008-08-25; First posted 2008-08-26 (Estimated); Last update posted 2011-09-30 (Estimated); Status verified 2011-09

CONDITIONS: Prostate Cancer
Keywords: vitamin D; prostate cancer; prostatectomy; pathology; immunohistochemistry
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator): vitamin D3 (400 IU/d)
  Interventions: Dietary Supplement: vitamin D3 (cholecalciferol)
- 2 (Active Comparator): vitamin D3 (10,000 IU/d)
  Interventions: Dietary Supplement: vitamin D3 (cholecalciferol)
- 3 (Active Comparator): vitamin D3 (40,000 IU/d)
  Interventions: Dietary Supplement: vitamin D3 (cholecalciferol)

INTERVENTIONS:
Dietary Supplement: vitamin D3 (cholecalciferol) — liquid vitamin D solution (vitamin D3 in ethanol) taken daily at one of three possible doses (400, 10000, or 40000 IU/d) for 4-6 weeks prior to radical prostatectomy

SUMMARY:
There is much interest in understanding the role that vitamin D3 (cholecalciferol) plays in various cancers, and in the prognosis of various cancers once they are discovered. The purpose of this study is to examine the effects of vitamin D on prostate cancer-associated lesions and on vitamin D metabolites in prostate tissue. We will give vitamin D3 to men when they are scheduled to have their prostate removed because of cancer. The men will take vitamin D at one of 3 doses for 4-6 weeks, until the surgery is performed. We will compare the prostate tissue taken from the men receiving the higher doses of vitamin D to tissue from men assigned to the lower doses. We expect to find that the prostate removed at surgery from men who received the high-dose vitamin D treatment will appear more normal, and less cancer like. In addition, we will measure vitamin D metabolites in the prostate to confirm that these did accumulate in the prostate to bring about the effects observed.

DETAILED DESCRIPTION:
Epidemiologic, laboratory, and clinical reports all suggest that vitamin D3 (cholecalciferol) plays a desirable role in the prevention and prognosis of prostate and other cancers. Prostate cancer cells possess both of the enzymes required to convert vitamin D to the active paracrine hormone, calcitriol. However, the dose-response relationship between serum levels of calcidiol (vitamin D status) and prostate tissue levels of calcidiol and calcitriol is yet to be defined. As a neoadjuvant, prior to radical prostatectomy (for 4-6 wk) vitamin D3 [400 IU (control group), 10,000 IU or 40,000 IU/day] will be given to 90 men randomized, double-blinded, 30 per dose. Immediately after surgery, the pathologist will obtain a few grams of prostate tissue, some of which will be used to assay calcidiol and calcitriol within prostate. From the embedded prostate, we will prepare immunohistochemically stained sections to characterize cellular responses and morphological changes. Our hypothesis is that vitamin D will increase intraprostate calcitriol concentration and thereby lower cellular proliferation (as judged by the markers MIB-1 and p27) in zones of Gleason pattern 3 prostate cancer and in pre-cancerous (PIN) lesions. We expect that our results will provide surrogate outcomes to justify larger trials of vitamin D for treatment of prostate cancer. This research has the potential to: 1. Provide direct evidence at the cellular level using clinical samples that vitamin D lowers cellular proliferation in prostate cancer, 2. Provide guidance about the serum calcidiol concentrations (and thereby vitamin D doses) that should be targeted for such studies, and 3. Eventually support other research directed at vitamin D as a primary prevention strategy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of a Gleason score 6 or 7 adenocarcinoma of the prostate biopsy
* Patient has elected to have a radical prostatectomy
* Patient is determined fit for surgery
* Normal renal and hepatic function
* Normal serum and urine calcium values
* Normal serum phosphate values
* Normal serum parathyroid hormone values
* Signed written informed consent

Exclusion Criteria:

* Prior use of neoadjuvant androgen deprivation therapy
* Prior use of 5 alpha reductase inhibitors (finasteride or dutasteride) in last 12 months
* Previous or concomitant anti-cancer therapy (chemotherapy, radiotherapy)
* Gleason score 8-10 adenocarcinoma as a biopsy diagnosis
* History of hypercalcemia/hypercalciuria
* History of renal disease
* History of sarcoidosis
* Vitamin D (cholecalciferol) supplement > 1000 IU/day
* Inability to comply with a study protocol

Ages: 30 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2008-09; Primary Completion 2012-02 (Estimated); Study Completion 2012-07 (Estimated)

PRIMARY OUTCOMES:
immunohistochemical markers of prostate pathology | end-of-study
intraprostate vitamin D metabolites | end-of-study

SECONDARY OUTCOMES:
calcium (serum and urine) | biweekly
parathyroid hormone (PTH) | baseline, final
prostate specific antigen (PSA) | baseline, final
creatinine (serum and urine) | biweekly
phosphate (serum) | biweekly
serum vitamin D metabolites | baseline, final

CONTACTS AND LOCATIONS:
Overall Officials: Reinhold Vieth, PhD, Principal Investigator — University of Toronto, Mount Sinai Hospital; Dennis Wagner, MSc, Study Director — University of Toronto, Mount Sinai Hospital; Theo van der Kwast, MD, PhD, FRCPC, Principal Investigator — University Health Network, Toronto; Neil Fleshner, MD, MPH, FRCSC, Principal Investigator — University Health Network, Toronto; Laurence Klotz, MD, FRCSC, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- University Health Network, Toronto, Ontario, Canada